CLINICAL TRIAL: NCT04154917
Title: Comparative Effectiveness of a Comprehensive, Patient-centered Hospital Discharge Planning Intervention (HOME) for Frail Older Adults: Feasibility Study for a Large Mixed-method Randomized Pragmatic Trial
Brief Title: Effectiveness of a Comprehensive Patient-centered Hospital Discharge Planning Intervention for Frail Older Adults
Acronym: HOME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Véronique Provencher, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 389430
Record Dates: First submitted 2019-10-28; First posted 2019-11-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Frail Older Adults
Keywords: Discharge planning; Frail older adults; Comprehensive approach; Patient-centered intervention

STUDY DESIGN:
Intervention Model Description: A feasibility study including a pragmatic, rater-blinded, mixed-method pilot RCT will be conducted over a 2 year-period to prepare for our large-scale planned study design. 72 frail older adults will be consecutively recruited from 2 acute care wards (geriatric and medicine units) in a hospital located in a semi-urban area (Sherbrooke, Quebec). Participants will be randomly assigned to receive HOME (experimental; n=36) or customary discharge planning (control; n=36). The number of participants is achievable within the time frame as, based the number of beds and average length of stay, approximately 1200 potential eligible patients are admitted yearly. This number (n=72) would make it possible to detect a large effect size, based on calculation for primary outcomes (α = 0.05; power = 80%) and the expected dropout rate (a ≈ 16-20%). Randomization will occur after baseline assessment using randomly generated numbers provided by a statistician not involved in data collection.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): HOME will be delivered by a community-based OT, who will be involved in the hospital discharge planning, trained by the PI. The HOME intervention comprises 4 phases: Phase 1 (in hospital): The clinician will focus on building a rapport with the patient and family members. Information will be gathered about the participant's home environment and functional ability. Phase 2 (± 5 days prior to expected discharge): Clinician will conduct a pre-discharge home assessment with patient and family to evaluate the environment, identify potential problems, and suggest appropriate ways to address them. Phase 3 (<1 week after discharge): Post-discharge home assessment will be conducted to provide additional in-home training and follow up on any of the patient's unmet needs. Phase 4 (2-4 weeks post-discharge): Follow-up telephone calls will be made to provide ongoing support to participant and family and encourage self-problem solving and independence.
  Interventions: Other: HOME
- Usual care (No Intervention): Usual care group will receive the customary discharge planning assessment by a different clinician (OT). During this assessment, according to usual care, information regarding the participants' ability to perform activities of daily living and regarding their home environment is gathered and used to plan for discharge. Usual care group will not receive an OT home assessment as this is not part of usual care. If the clinician identifies a potential need for assistive equipment and home modification needs, patients will be referred to community-based homecare services as is the current practice, and a home visit may be performed following discharge, typically after an lengthy wait (weeks, months) for service.

INTERVENTIONS:
Other: HOME — HOME's focus is on the person's functional ability, safety and transition from hospital to home. HOME will be delivered by a community-based clinician (OT who will be involved in the hospital discharge planning) trained by the PI. Training will include two sessions covering assessment of functional ability, goal setting and home safety. The clinician will keep a record of recommendations provided, length of home visit and any adverse events during the intervention. Twice over the course of the study, the PI leader will observe the clinician conducting HOME interventions to assess adherence to the study protocol using a fidelity checklist. The HOME intervention comprises 4 phases, which are described in the arms section.
  Arms: Experimental

SUMMARY:
A large number of frail older adults have difficulty performing activities of daily living and resuming former roles in the months following hospital discharge. This increases the risk of unplanned hospital readmissions and emergency visits after they return home. Comprehensive, patient-centered discharge planning has been reported to improve older adults' ability to perform activities of daily living and to reduce readmission rates after hospital discharge. However, to our knowledge, no evidence-based discharge protocol is routinely used in Canada with the frail population. An innovative discharge planning intervention called "HOME" was recently developed in Australia, which includes: 1) hospital based partnership with patient and family to establish goal setting and problem solving; 2) pre-discharge home assessment to address safety issues and problems with patient and family; 3) post-discharge home assessment and in-home training to address unmet needs; and 4) follow-up telephone calls to provide ongoing support to patient and family. A Canadian version of HOME has been developed. This will be followed by a large trial to investigate if this intervention increases functioning in daily life activities and decreases hospital and emergency readmissions for frail patients who are discharged home. Our proposed study is a preliminary and necessary step to identify problems that may arise during this large trial and address them proactively. If proven beneficial, the Canadian version of HOME would be an appropriate, applicable and acceptable intervention to improve patients' experiences and outcomes as well as change health practice surroundings discharge planning with frail older adults.

DETAILED DESCRIPTION:
Up to 31% of frail patients are readmitted to hospital within 30 days post-discharge. Unmet needs related to new difficulties in performing activities of daily living (ADL) upon returning home increase their risk of readmission. Comprehensive, patient-centered discharge planning has been reported to improve older adults' ability to perform ADL and to reduce readmission rates. To our knowledge, no such evidence-based discharge protocol is routinely used in Canada with the frail population.

An innovative discharge planning protocol called "HOME" was recently developed in Australia and a randomized controlled trial (RCT) was conducted in a large sample of older adults in this country. The HOME intervention includes: 1-hospital-based partnership with patient and family to establish goal setting and problem solving; 2-pre-discharge home assessment to address safety issues and problems with patient and family; 3-post-discharge home assessment training to address unmet needs; and 4-Follow-up telephone calls to provide ongoing support to patient and family. Using the HOME protocol in a real-world Canadian context is expected to yield positive functional and clinical outcomes for this population. This hypothesis needs to be verified through a full-scale pragmatic mixed-method (qualitative and quantitative) RCT. This innovative method supports the integration of research into care and increase understanding of the results. Given the changes we are making to the Australian design and the different context in which the research will be done, a feasibility study will first be conducted to help circumvent problems that may arise during the full-scale RCT. Thus this study aims to assess the feasibility of conducting a fully powered multi-site, pragmatic, mixed-method RCT that will evaluate the comparative effectiveness of a Canadian version of HOME with respect to (a) functional outcomes: independence in ADL and functional goal attainment; and (b) clinical outcomes: unplanned hospital readmissions and emergency department visits.

A pragmatic pilot RCT using a rater-blinded mixed-method design will be conducted over a 2-year period. Seventy-two frail hospitalized older adults will be consecutively recruited in Sherbrooke (Quebec). Participants will be randomly allocated to the intervention group (HOME) or the control group (customary in-hospital care). Feasibility data, including recruitment and retention rates, will be collected. Quantitative methods will be used to explore the effect of the HOME intervention on (a) functional outcomes, measured by the Functional Autonomy Measurement System and the Goal Attainment Scale, and (b) clinical outcomes based on medical chart data reviews. A qualitative method embedded in the RCT will be used to explore how the intervention is experienced by clinicians, patients and families to plan further refinements. Measures will be taken at baseline, 1 and 3 months post-discharge.

With the participation of the Australian research team and a network of patient-caregiver representatives, clinicians, and key policy makers (e.g., Quebec Ministry of Health), this study will provide clinically-relevant results to support the full-scale RCT. By providing evidence on the effectiveness, benefits and potential drawbacks in a real-world context of the two options (HOME vs customary care), findings from this RCT will help stakeholders make decisions about the best way of delivering discharge planning care for frail patients.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* have mild cognitive impairment (MoCA range score: 20-26)
* are expected to return to live in the community after discharge
* are conversant in French or English
* expected hospital stay should be > or = 5 days
* should have a family member who agrees to participate in the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Functional autonomy measure (SMAF) at 1 and 3 months after discharge | in the hospital at baseline (T1); at the patient's home 1 month (T2) and 3 months (T3) after discharge
  SMAF is a 29-item scale based on the WHO Classification of Disabilities. It measures functional ability in five areas: ADL (7 items), mobility (6 items), communication (3 items), mental functions (5 items), and IADL (8 items). Each item is scored from 0 (independent) to 3 (dependent) for a maximum total score of 87. A change of ≥5 points is considered clinically significant.
Change in Unplanned hospital readmissions at 1 and 3 months after discharge | 1 and 3 months post-discharge
  Unplanned hospital readmissions will be collected through chart reviews via the Ariane database. Readmissions will be classified as unplanned based on the medical ICD010-OMS classification ("avoidable incidents")

SECONDARY OUTCOMES:
Change from baseline Goal attainment scaling (GSA) at 3 months after discharge | from baseline to 3 months post discharge
  GAS is a personalized outcome measure involving i) setting goals according to one's own needs prior to the start of the intervention, ii) implementing the intervention, and iii) evaluating progress following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Provencher, Principal Investigator — Université de Sherbrooke
Locations (1):
- CIUSSS de l'Estrie CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No